CLINICAL TRIAL: NCT06386614
Title: The Second Hospital of Dalian Medical University
Brief Title: Effect of Frontal Transcranial Direct Current Stimulation on BDNF in Stroke Patients With Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BDNF
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- common group routine training (Sham Comparator): Conventional rehabilitation
  Interventions: Other: Routine treatment
- tDCS group (Experimental): Conventional rehabilitation plus TDCS treatment
  Interventions: Other: Routine treatment; Other: Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Routine treatment — Both groups were given routine treatment
  Other Names: Routine medical treatment; basic rehabilitation training; individualized cognitive training
Other: Transcranial Direct Current Stimulation — The common group routine training used sham TDCS stimulation, and the experimental group used real TDCS stimulation
  Arms: tDCS group

SUMMARY:
The purpose of the clinical trial is to find a treatment for stroke patients with cognitive impairment, and the main questions it aims to answer are:

* [Search for effective treatments of cognitive impairment after stroke]
* [explore the relationship between BDNF level and cognitive function] Participants will receive conventional treatment, tDCS treatment, .And then compare cognitive function and BDNF level

DETAILED DESCRIPTION:
1. To study the therapeutic effect of transcranial direct current stimulation (tDCS) on post-stroke cognitive impairment (PSCI) by evaluating cognitive function and detecting plasma brain-derived neurotrophic factor (BDNF).
2. To explore the correlation between plasma BDNF level and cognitive function in patients with PSCI.

ELIGIBILITY:
Inclusion Criteria:

* (1)Stroke patients with CT or MRI imaging evidence, among which ischemic stroke met the diagnostic criteria of Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018, and cerebral hemorrhage diseases met the diagnostic criteria of Chinese Guidelines for the Diagnosis and Treatment of Cerebral hemorrhage 2019; (2) There are symptoms related to cognitive dysfunction; Cognitive dysfunction was assessed by rehabilitation physicians. According to the MoCA evaluation standard,MoCA score ≤26 points; according to the MMSE evaluation standard, illiteracy score ≤17 points; primary school education level ≤20 points; secondary school education (including secondary school) level ≤22 points; college education (including junior college) level ≤23 points; (3)Age range 40-80 years old; (4) no obvious aphasia, speech expression and attention can cooperate with the completion of evaluation and treatment; (5)The patient or the patient's family members read and agree to sign the informed consent.

Exclusion Criteria:

* (1) Patients with severe diseases, such as malignant arrhythmia, acute myocardial infarction and acute heart failure, who cannot tolerate rehabilitation treatment; (2) Patients with untreated intracranial aneurysms, severe epilepsy, and intracranial metals who cannot receive tDCS treatment; (3) Non-PSCI patients with cognitive impairment, including patients with cognitive impairment left over from previous stroke and other organ disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
BDNF | 2 weeks
  Plasma BDNF was determined by elisa

SECONDARY OUTCOMES:
Cognitive function level | 2 weeks
  Score of Mini-Mental State Examination(MMSE) and Montreal Cognitive Assessment(MoCA)
Executive function level | 2 weeks
  core of The Frontal Assessment Battery（FAB）
Memory function level | 2 weeks
  Score of Rivermead Behavioral Memory Test（RBMT）

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Jiang, Study Director — Department of Rehabilitation Medicine, the Second Hospital of Dalian Medical University
Locations (2):
- China (2):
  - Department of Rehabilitation Medicine, the Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Lily, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No